CLINICAL TRIAL: NCT02300233
Title: The COMPASS Study: A Randomized, Double-Blind, Placebo-Controlled Phase 3 Study of ISIS 304801 Administered Subcutaneously to Patients With Hypertriglyceridemia
Brief Title: The COMPASS Study: A Study of Volanesorsen (Formally ISIS-APOCIIIRx) in Patients With Hypertriglyceridemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Collaborators: Akcea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ISIS 304801-CS16; 2014-003434-93 (EudraCT Number)
Record Dates: First submitted 2014-11-20; First posted 2014-11-24 (Estimated); Results first posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-03

CONDITIONS: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia | interventions — ISIS 304801

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Volanesorsen-matching placebo administered subcutaneously once-weekly for 26 weeks.
  Interventions: Drug: Placebo
- Volanesorsen 300 mg weekly (Experimental): Volanesorsen 300 mg administered subcutaneously once-weekly for 26 weeks.
  Interventions: Drug: Volanesorsen
- Volanesorsen 300 mg biweekly, post Week 13 (Experimental): Volanesorsen 300 mg administered subcutaneously once-weekly for 13 weeks, then bi-weekly for 13 weeks.
  Interventions: Drug: Volanesorsen

INTERVENTIONS:
Drug: Volanesorsen — 300 mg volanesorsen administered subcutaneously once-weekly for 26 weeks.
  Other Names: ISIS 304801
  Arms: Volanesorsen 300 mg biweekly, post Week 13; Volanesorsen 300 mg weekly
Drug: Placebo — Volanesorsen-matching placebo administered subcutaneously once-weekly for 26 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of volanesorsen given for 26 weeks in participants with Hypertriglyceridemia.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) ≤ 45 kg/m2
2. Fasting Triglycerides (TG) ≥ 500 mg/dL (≥ 5.7 mmol/L) at Screening.
3. If on statin or fibrate, participants must be on stable, labeled dose for at least 3 months prior to screening. Participants not receiving these drugs within 4 weeks prior to screening are also eligible.

Exclusion Criteria:

1. Type 1 diabetes mellitus
2. Newly diagnosed type 2 diabetes mellitus (within 12 weeks of screening) or HbA1c ≥ 9.0% at Screening
3. Acute pancreatitis within 3 months of screening
4. Acute Coronary Syndrome within 6 months of screening
5. Major surgery within 3 months of screening
6. Prior exposure to ISIS 304801
7. Have any other conditions in the opinion of the investigator which could interfere with the participant participating in or completing the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2015-02-05 (Actual); Primary Completion 2016-07-27 (Actual); Study Completion 2017-01-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (44):
- United States (28):
  - IONIS Investigative Site, Encinitas, California
  - IONIS Investigative Site, San Francisco, California
  - IONIS Investigative Site, Boca Raton, Florida
  - IONIS Investigative Site, Miami, Florida
  - IONIS Investigative Site, Sterling, Illinois
  - IONIS Investigative Site, Kansas City, Kansas
  - IONIS Investigative Site, Salisbury, Maryland
  - IONIS Investigative Site, Towson, Maryland
  - IONIS Investigative Site, Boston, Massachusetts
  - IONIS Investigative Site, Grandville, Michigan
  - IONIS Investigative Site, North Massapequa, New York
  - IONIS Investigative Site, Benson, North Carolina
  - IONIS Investigative Site, Chapel Hill, North Carolina
  - IONIS Investigative Site, Farmville, North Carolina
  - IONIS Investigative Site, Greenville, North Carolina
  - IONIS Investigative Site, Morrisville, North Carolina
  - IONIS Investigative Site, Raleigh, North Carolina
  - IONIS Investigative Site, Wilson, North Carolina
  - IONIS Investigative Site, Cincinnati, Ohio
  - IONIS Investigative Site, Kettering, Ohio
  - IONIS Investigative Site, Marion, Ohio
  - IONIS Investigative Site, Oklahoma City, Oklahoma
  - IONIS Investigative Site, Portland, Oregon
  - IONIS Investigative Site, Providence, Rhode Island
  - IONIS Investigative Site, Houston, Texas
  - IONIS Investigative Site, Salt Lake City, Utah
  - IONIS Investigative Site, Norfolk, Virginia
  - IONIS Investigative Site, Seattle, Washington
- Canada (4):
  - IONIS Investigative Site, Vancouver, British Columbia
  - IONIS Investigative Site, London, Ontario
  - IONIS Investigative Site, Chicoutimi, Quebec
  - IONIS Investigative Site, Sainte-Foy, Quebec
- France (4):
  - IONIS Investigative Site, Dijon
  - IONIS Investigative Site, Marseille
  - IONIS Investigative Site, Paris
  - IONIS Investigative Site, Saint-Herblain
- Germany (3):
  - IONIS Investigative Site, Cologne, North Rhine-Westphalia
  - IONIS Investigative Site, Berlin
  - IONIS Investigative Site, Dresden
- Netherlands (3):
  - IONIS Investigative Site, Amsterdam, North Holland
  - IONIS Investigative Site, Rotterdam, South Holland
  - IONIS Investigative Site, Utrecht
- United Kingdom (2):
  - IONIS Investigative Site, Manchester
  - IONIS Investigative Site, Peterborough

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prohaska TA, Alexander VJ, Karwatowska-Prokopczuk E, Tami J, Xia S, Witztum JL, Tsimikas S. APOC3 inhibition with volanesorsen reduces hepatic steatosis in patients with severe hypertriglyceridemia. J Clin Lipidol. 2023 May-Jun;17(3):406-411. doi: 10.1016/j.jacl.2023.04.007. Epub 2023 Apr 27. PMID 37164837
- [Derived] Gouni-Berthold I, Alexander VJ, Yang Q, Hurh E, Steinhagen-Thiessen E, Moriarty PM, Hughes SG, Gaudet D, Hegele RA, O'Dea LSL, Stroes ESG, Tsimikas S, Witztum JL; COMPASS study group. Efficacy and safety of volanesorsen in patients with multifactorial chylomicronaemia (COMPASS): a multicentre, double-blind, randomised, placebo-controlled, phase 3 trial. Lancet Diabetes Endocrinol. 2021 May;9(5):264-275. doi: 10.1016/S2213-8587(21)00046-2. Epub 2021 Mar 30. PMID 33798466

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 114 participants were randomized at multiple study centers worldwide.
Pre-assignment Details: 114 participants were randomized, and 113 received study drug. One patient was randomized, but discontinued before dosing, and thus included only in the volanesorsen Total (Not public) column. The study included a ≤ 8-week screening period (including a diet-stabilization period), a 26-week treatment period, and a 13-week post-treatment evaluation period.
Period: Overall Study
Arm/Group | Placebo | Volanesorsen 300 mg Weekly | Volanesorsen 300 mg Biweekly, Post Week 13
Started | 38 | 25 | 50
Completed (Completed here refers to participants who completed the study treatment.) | 34 | 24 | 27
Not Completed | 4 | 1 | 23
Not completed — Adverse Event or Serious Adverse Event | 3 | 1 | 14
Not completed — Withdrawal by Subject | 1 | 0 | 3
Not completed — Investigator Judgement | 0 | 0 | 1
Not completed — Reason Not Specified | 0 | 0 | 5

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all participants who were randomized, received at least one dose of study drug, and had a baseline triglycerides (TG) assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Volanesorsen 300 mg Weekly | Volanesorsen 300 mg Biweekly, Post Week 13 | Total
Number analyzed (Participants) | 38 | 25 | 50 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (10) | 50 (9) | 51 (11) | 51 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 14 | 27
  Male | 30 | 20 | 36 | 86
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 37 | 24 | 50 | 111
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 33 | 25 | 47 | 105
  Asian | 3 | 0 | 1 | 4
  American Indian or Alaskan Native | 0 | 0 | 1 | 1
  Other Race | 1 | 0 | 1 | 2
  Multiple | 1 | 0 | 0 | 1
Fasting Triglycerides [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] | 1414 (1253) | 1046 (560) | 1251 (838) | 1261 (955)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Fasting Triglycerides (TG) From Baseline to Month 3
Time Frame: Baseline to 3 months
Population: The full analysis set (FAS) included all participants who were randomized, received at least one dose of study drug, and had a baseline TG assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Groups:
- Volanesorsen Total: Volanesorsen 300 mg administered subcutaneously once-weekly for 26 weeks; or once-weekly for 13 weeks, then bi-weekly for 13 weeks.
Arm/Group | Placebo | Volanesorsen Total
Number analyzed (Participants) | 38 | 75
percent change | -0.9 [-13.9 to 12.2] | -71.2 [-79.3 to -63.2]
Statistical Analysis 1: Comparison: Placebo vs Volanesorsen Total; Test type: Superiority; p < 0.0001, ANCOVA; Difference in Least Squares Mean (LSM) = -70.3, 95% CI 2-sided [-85.4 to -55.3]

2. Secondary Outcome: Absolute Change in Fasting TG From Baseline to Month 3
Time Frame: Baseline to 3 months
Population: The FAS included all participants who were randomized, received at least one dose of study drug, and had a baseline TG assessment. Volanesorsen 300 mg biweekly group includes patients who received weekly dosing in first 13 weeks, and then bi-weekly for 13 weeks. For month 3 assessments, the results were combined since all patients were on weekly dosing. And for month 6 assessments, the results were split to show the results in each dosing group.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Placebo | Volanesorsen Total
Number analyzed (Participants) | 38 | 75
mg/dL | 74 [-138 to 285] | -869 [-1018 to -720]
Statistical Analysis 1: Comparison: Placebo vs Volanesorsen Total; Test type: Superiority; p < 0.0001, ANCOVA; Difference in LSM = -943, 95% CI 2-sided [-1197 to -689]

3. Secondary Outcome: Treatment Response Rate Defined as Participants With Fasting TG ≥ 40% Reduction From Baseline at Month 3
Time Frame: Baseline to 3 months
Population: The FAS included all participants who were randomized, received at least one dose of study drug, and had a baseline TG assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Volanesorsen Total
Number analyzed (Participants) | 38 | 75
Participants | 5 | 65
Statistical Analysis 1: Comparison: Placebo vs Volanesorsen Total; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 96.02, 95% CI 2-sided [19.71 to 467.79]

4. Secondary Outcome: Percent Change in High-density Lipoprotein-cholesterol (HDL-C) From Baseline
Time Frame: Baseline to 3 months
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Volanesorsen Total
Number analyzed (Participants) | 38 | 75
percent change | 4.4 [-5.2 to 14.0] | 61.2 [54.2 to 68.3]
Statistical Analysis 1: Comparison: Placebo vs Volanesorsen Total; Test type: Superiority; p < 0.0001, ANCOVA; Difference in LSM = 56.8, 95% CI 2-sided [45.1 to 68.6]

5. Secondary Outcome: Treatment Response Rate Defined as Participants With Fasting TG < 150 mg/dL Reduction From Baseline at Month 3
Description: mg/dL = milligrams per deciliter
Time Frame: Baseline to 3 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Volanesorsen Total
Number analyzed (Participants) | 38 | 75
Participants | 0 | 11
Statistical Analysis 1: Comparison: Placebo vs Volanesorsen Total; Test type: Superiority; p = 0.0474, Regression, Logistic; Odds Ratio (OR) = 14.93, 95% CI 2-sided [1.03 to 215.88]

6. Secondary Outcome: Change From Baseline in Homeostasis Model Assessment-estimated Insulin Resistance (HOMA-IR)
Description: HOMA-IR was calculated using the following formula: fasting insulin micro-international units per millimeter (μIU/mL) x fasting glucose mg/dL]/405. A negative change from baseline indicates improvement; a positive change from baseline indicates worsening.
Time Frame: Baseline to 3 and 6 months
Population: The FAS included all participants who were randomized, received at least one dose of study drug, and had a baseline TG assessment. Number analyzed were the participants evaluated at the given time point.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Placebo | Volanesorsen 300 mg Weekly | Volanesorsen 300 mg Biweekly, Post Week 13
Number analyzed (Participants) | 38 | 25 | 50
score
  Month 3: number analyzed (Participants) | 36 | 24 | 42
  Month 3 | -0.29 (3.12) | 1.53 (4.89) | -0.45 (4.97)
  Month 6: number analyzed (Participants) | 35 | 24 | 38
  Month 6 | -0.37 (3.18) | 1.54 (7.69) | 0.56 (2.97)

7. Secondary Outcome: Change From Baseline in Glycated Hemoglobin (HbA1c) in Type 2 Diabetes Mellitus (T2DM) Participants
Time Frame: Baseline to 3 and 6 months
Population: The FAS included all participants who were randomized, received at least one dose of study drug, and had a baseline TG assessment. Number analyzed were the T2DM participants evaluated at the given time point.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Placebo | Volanesorsen 300 mg Weekly | Volanesorsen 300 mg Biweekly, Post Week 13
Number analyzed (Participants) | 14 | 9 | 21
percentage
  Month 3: number analyzed (Participants) | 13 | 9 | 21
  Month 3 | -0.0 (0.5) | 0.4 (0.6) | 0.1 (0.5)
  Month 6: number analyzed (Participants) | 12 | 9 | 19
  Month 6 | -0.2 (0.6) | 0.8 (0.9) | 0.3 (0.9)

ADVERSE EVENTS:
Time Frame: Up to approximately 39 weeks.
Description: The safety set included all randomized participants who received at least one dose of study drug.
Arm/Group | Placebo | Volanesorsen 300 mg Weekly | Volanesorsen 300 mg Biweekly, Post Week 13
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/25 | 0/50
Serious Adverse Events (participants affected / at risk) | 4/38 | 2/25 | 6/50
Other Adverse Events (participants affected / at risk) | 31/38 | 24/25 | 49/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=38) | Volanesorsen 300 mg Weekly (N=25) | Volanesorsen 300 mg Biweekly, Post Week 13 (N=50)
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 2 | 1 | 0
Pancreatitis relapsing (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Serum sickness (Immune system disorders) | 0 | 0 | 1
Pancreas infection (Infections and infestations) | 1 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=38) | Volanesorsen 300 mg Weekly (N=25) | Volanesorsen 300 mg Biweekly, Post Week 13 (N=50)
Injection site erythema (General disorders) | 2 | 23 | 38
Injection site pain (General disorders) | 2 | 10 | 29
Injection site swelling (General disorders) | 1 | 12 | 24
Injection site pruritus (General disorders) | 0 | 10 | 17
Injection site discolouration (General disorders) | 0 | 12 | 11
Injection site induration (General disorders) | 2 | 7 | 11
Injection site discomfort (General disorders) | 1 | 2 | 11
Fatigue (General disorders) | 4 | 2 | 7
Injection site bruising (General disorders) | 1 | 1 | 10
Injection site rash (General disorders) | 0 | 3 | 6
Pyrexia (General disorders) | 2 | 2 | 5
Injection site reaction (General disorders) | 0 | 4 | 4
Injection site warmth (General disorders) | 0 | 2 | 6
Asthenia (General disorders) | 2 | 3 | 2
Injection site haemorrhage (General disorders) | 0 | 2 | 5
Injection site hypoaesthesia (General disorders) | 0 | 1 | 5
Injection site inflammation (General disorders) | 1 | 2 | 2
Pain (General disorders) | 2 | 0 | 2
Injection site mass (General disorders) | 0 | 2 | 1
Injection site oedema (General disorders) | 0 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 4 | 5 | 5
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 9
Nausea (Gastrointestinal disorders) | 1 | 1 | 6
Vomiting (Gastrointestinal disorders) | 1 | 1 | 4
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 3
Nasopharyngitis (Infections and infestations) | 5 | 8 | 4
Bronchitis (Infections and infestations) | 3 | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 2
Urinary tract infection (Infections and infestations) | 2 | 2 | 0
Influenza (Infections and infestations) | 2 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 4
Red blood cell sedimentation rate increased (Investigations) | 4 | 6 | 5
C-reactive protein increased (Investigations) | 0 | 3 | 5
Low density lipoprotein increased (Investigations) | 0 | 3 | 4
Platelet count decreased (Investigations) | 2 | 1 | 2
Hepatic enzyme increased (Investigations) | 0 | 1 | 3
Blood creatinine increased (Investigations) | 0 | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2 | 8
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 3
Gout (Metabolism and nutrition disorders) | 2 | 1 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 0
Headache (Nervous system disorders) | 4 | 2 | 5
Dizziness (Nervous system disorders) | 2 | 2 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Depression (Psychiatric disorders) | 0 | 2 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 2 | 1
Albuminuria (Renal and urinary disorders) | 0 | 2 | 1
Hot flush (Vascular disorders) | 2 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes